CLINICAL TRIAL: NCT03929302
Title: Brain Energy Metabolism and Sleep in Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As the study involved recruitment of at risk population such as Alzheimer's disease, the study was terminated due to COVID situation/
Sponsor: The University of Texas at Dallas (Other)
Collaborators: Texas A & M University Baylor College Of Dentistry (Other); University of Texas, Southwestern Medical Center at Dallas (Other)
Responsible Party: Principal Investigator, Sandra Chapman, PhD, Founder and Chief Director, Center for BrainHealth® Dee Wyly Distinguished University Professor, The University of Texas at Dallas
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 18-73
Record Dates: First submitted 2019-03-12; First posted 2019-04-26 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Cognitive Change; Energy Metabolism; Sleep Disturbance
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Cognitively normal adults group (Active Comparator): A group of cognitively normal adults will be included to investigate whether MyTAP oral airway management with a mouth shield improves sleep and cognition.
  Interventions: Device: MyTAP oral appliance plus mouth shield
- Mild Cognitive Impairment (MCI) group (Active Comparator): A group of MCI will be included to investigate whether MyTAP oral airway management with a mouth shield improves sleep and cognition.
  Interventions: Device: MyTAP oral appliance plus mouth shield
- Alzheimer's Disease group (Active Comparator): A group of AD will be included to investigate whether MyTAP oral airway management with a mouth shield improves sleep and cognition.
  Interventions: Device: MyTAP oral appliance plus mouth shield

INTERVENTIONS:
Device: MyTAP oral appliance plus mouth shield — The midline traction oral appliance (MyTAP, AMI Inc., Dallas, Texas) is currently marketed as a medical device to treat snoring and obstructive sleep apnea and is FDA cleared will be used in all the three arms.

SUMMARY:
The three primary goals of this pilot will be followed by a secondary goal to test if dental intervention improves brain health in terms of sleep and cognition. The primary and secondary goals are

1. Explore the ratios of brain energy (ATP/PCr, Pi/PCr) and phospholipids (PME/PDE) metabolites as measured by magnetic resonance spectroscopy at 7 Tesla, and compare the differences in them with the performance of episodic memory, attention, language, and executive functions (abstraction, reasoning, verbal fluency, working memory) in three groups: cognitively normal adults, mild cognitive impairment (MCI) and Alzheimer's disease (AD).
2. Investigate the differences in sleep patterns measured by the ratio sleep quality index (Stable/ Unstable sleep) in cognitively normal adults, MCI and AD and its relation to the performance of episodic memory, attention, language, and executive functions (abstraction, reasoning, verbal fluency, working memory) in three groups.
3. Investigate the differences in the variations of two genes, APOE-E4 and ABCA7, in relationship to the changes in the brain energy metabolites and its relation to the performance of episodic memory, attention, language, and executive functions (abstraction, reasoning, verbal fluency, working memory) in those with cognitively normal adults, MCI and AD.
4. Investigate if dental intervention improves sleep patterns and overall cognitive behavior in the three cohorts.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is rapidly progressing in the elder population and the pathophysiological changes in the brain start at least 1-2 decades before the disease onset. During this period of slow progression, individuals may notice subtle changes in the memory and this subset of the population is termed as Mild Cognitive Impairment (MCI). MCI is a pre-clinical stage of Alzheimer's disease (AD) in which individuals have memory complaints but are functionally independent and not yet clinically diagnosed with dementia. New modalities for potential identification of the progression of the disease, include different biomarkers, state-of-the-art technologies like sleep tracking and magnetic resonance spectroscopy (MRS) may provide additional, essential tools to facilitate early detection of disease, which may allow for earlier intervention and provide a potential gauge for a response to treatment.

The first goal of this research project aims to understand the variations in the brain energy and phospholipid metabolites as measured by magnetic resonance spectroscopy at 7 Tesla across three groups: cognitively healthy adults, MCI, and AD. The brain requires a lot of energy in the form of adenosine triphosphate (ATP) to support the neuronal activity, and it has a rich source of phospholipids to maintain biological functions. Therefore, abnormalities in the mechanism of energy supply and phospholipids can affect a wide range of function in the neuronal cells. Previous literature using 18FDG PET scan has shown impairments in brain glucose metabolism associated with cognitive decline in MCI even before the individual presents with clinically apparent cognitive dysfunction. Thus, measuring the ratio of energy metabolites ATP-to-PCr (ATP/PCr) and Pi-to-PCr (Pi/PCr) offers a promising way to predict the active status of the resting brain.

Additionally, the levels of phospholipids start to decrease by the age of twenty (20), and more pronounced decline is noticed after the age of 80 years. Thus, aging and diseased brains are more susceptible to the changes in the levels of phospholipids metabolites which can lead to neurodegenerative disorders. Two classes of phospholipid metabolites that can be studied using 31P MRS are phosphomonoesters (PMEs) and phosphodiesterase (PDEs). PMEs are the essential building blocks for cell/neuronal membrane synthesis whereas PDEs are the metabolites from the breakdown of the cell/neuronal phospholipids membrane. A higher ratio of PMEs-to-PDEs can, therefore, reflect as an improvement in brain health leading to neurogenesis, with the opposite suggesting neurodegeneration. Thus, 31P MRS has opened a window to measure various neurochemical metabolites non-invasively, which could provide detailed information about important high-energy phosphate metabolites, as well as phospholipid metabolites in real time. 7T Ultra-high magnetic field MRI scanner, which is now increasingly accessible worldwide and enables fast and accurate BEM measurement, may provide a comprehensive approach for aiding in the diagnosis of the neurodegenerative process from cognitively normal adults to MCI and AD and also monitoring the treatment responses to newer drugs.

Secondly, disturbance in sleep patterns can impact the brain's energy metabolism by altering the ratio of brain energy and phospholipid metabolites, thereby causing impaired brain cognitive functions. Aging is a significant moderator of sleep quality and may affect non-REM slow wave sleep (SWS), which facilitates the clearance of toxic material like amyloid protein. Stable sleep helps restore the neurobiological and neurophysiological responses about energy requirements impacting the changes in the concentration of brain energy and phospholipid metabolism. Currently, data are lacking regarding the relationship between sleep, brain energy requirement and its effect on the performance of cognitive domains to healthy aging, MCI, and AD.

Thirdly, BEM is regulated by specific genes that support the continuous energy requirements for the electrical activity of the brain. Hence in this research, we are interested in investigating the effect of two genes APOE ε4 and ABCA7 on brain energy and phospholipids metabolites in the three groups. It is essential to understand this connection as genes regulate the synthesis of appropriate protein/enzymes like ABCA7 transporter protein for glucose metabolism leading to energy production.

Finally, based on an "improving sleep first hypothesis," a dental intervention (MyTAP; midline traction oral appliance (OA) therapy will be offered to participants presenting with abnormal sleep and upper airway obstruction parameters. Therapeutic response to attenuate upper airway obstruction in sleep by using continuous positive airway pressure (CPAP) was shown also to improve cognitive functioning in AD patients with OSA. In most cases, upper airway obstruction can also be acutely corrected using a simple fitted, clinically proven, FDA-cleared midline traction design oral appliance to restore sleep quality and possibly improve cognition and 'normalize' BEM. There are currently no reports on the efficacy of oral appliance therapy to improve daytime sleepiness, objective sleep measures and cognitive function in patients with MCI or AD. The MyTAP is similar to other midline traction design oral appliances which have been in clinical use for over 20 years without any serious adverse effects in treating patients with primary snoring to severe sleep apnea The MyTAP oral appliance will be used in accordance with its indications for use and FDA-approved labeling. The safety and efficacy of the midline traction oral appliance have already been published. As per FDA cleared label MyTAP® OA family of intra-oral devices are intended for the treatment of night-time snoring and mild to moderate obstructive sleep apnea in patients 18 years of age or older.

All eligible participant agreeing to sign the consent form and participate in the study will be divided into 3 groups - Cognitively Normal Adults, MCI and AD based on Mini Mental Status Examination (MMSE) and California Verbal Learning Task (CVLT). All participants will initially undergo the mandatory set of study procedures for neurocognitive testing, genetic testing, MRS scan and sleep assessment. Interested participants in all the 3 groups, presenting with abnormal sleep and upper airway obstruction parameters during the sleep assessment will then be offered the optional therapeutic intervention Intraoral anti-snoring device for snoring and obstructive sleep apnea for three months.

ELIGIBILITY:
Inclusion Criteria: Eligible participants will be:

* Ages 55-85 years
* At least 12 years of education
* Right hand dominant
* With or without minor memory complaints (those with a diagnosis of Alzheimer's disease,
* Participants who can safely have an MRS scan
* Have motor abilities including the use of the right arm and hand for neuropsychological testing.
* Able to speak, read, and comprehend English fluently
* Non-pregnant, and not on Hormone replacement therapy

Exclusion criteria will be:

* Pregnancy
* Use of Hormone Replacement therapy
* Less than 12 years of education
* Left hand dominant
* Unable to speak, read and write English fluently (Testing and training material are validated in English).
* Neurological Disorders, e.g., stroke, brain tumor, cerebral hemorrhage.
* Autoimmune disorders like fibromyalgia, systemic lupus erythematosus (SLE), Multiple sclerosis and rheumatoid arthritis.
* Metabolic diseases such as diabetes mellitus, thyroid disorders that are not currently managed by a physician
* Psychiatric disorders such as bipolar disorder, major depressive disorder, pervasive developmental disorder, schizophrenia, anxiety disorder.
* Current drug or alcohol abuse
* Head injuries with an Ohio State University TBI Identification (Short Form) score greater than 3.
* Cancer treated with radiation and/or chemotherapy
* General anesthesia within the prior six months
* Uncorrected vision and hearing problems.
* Active pain requiring treatment
* BMI ≥35
* Previously diagnosed sleep disorders
* Known chronic obstructive pulmonary disease(COPD)
* Exclusion for imaging criteria (includes the following, or any other concerns by the AIRC staff)

  * Permanent Makeup.
  * Exclusions for metal safety include questionable ferrous implants, bullets, BB's, shrapnel,
  * Medical devices which are unsafe in MRI.
  * Hearing aid that cannot be removed.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for BrainHealth, The University of Texas at Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 248 participants were screened for eligibility criteria, of which 41 consented by signing the informed consent to participate in the study in three arms: cognitively normal, mild cognitive impairment, and Alzheimer's disease.
Groups:
- Cognitively Normal Adults Group; Mild Cognitive Impairment (MCI) Group; Alzheimer's Disease Group: Part A-The basic science of the relationship of sleep abnormalities, genes, brain energy metabolites variables with cognitive performance will be explored.
  Part B- A sample of the group will be included to investigate whether MyTAP oral airway management with a mouth shield improves sleep and cognition.
Period: Neurocognitive and MRS Testing
Arm/Group | Cognitively Normal Adults Group | Mild Cognitive Impairment (MCI) Group | Alzheimer's Disease Group
Started (Part A enrollment) | 15 | 15 | 11
Completed | 15 | 15 | 11
Not Completed | 0 | 0 | 0
Period: Intervention - myTAP Mouth Shield
Arm/Group | Cognitively Normal Adults Group | Mild Cognitive Impairment (MCI) Group | Alzheimer's Disease Group
Started | 15 | 15 | 11
Completed | 7 | 7 | 6
Not Completed | 8 | 8 | 5
Not completed — Withdrawal by Subject | 5 | 8 | 4
Not completed — Time constraints | 3 | 0 | 0
Not completed — Device didnot fit | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: At baseline, a total of 41 participants were enrolled in three respective groups.
  is 32 of which only 22 participant data were useable. The reason for attrition is due to either noncompliance of training or unable to use the MRI data due to movement.
Groups:
- Mild Cognitive Impairment Group; Alzheimer's Disease Group: Part A-The basic science of the relationship of sleep abnormalities, genes, brain energy metabolites variables with cognitive performance will be explored.
  Part B- A sample of the group will be included to investigate whether MyTAP oral airway management with a mouth shield improves sleep and cognition.
- Total: Total of all reporting groups
Arm/Group | Cognitively Normal Adults Group | Mild Cognitive Impairment Group | Alzheimer's Disease Group | Total
Number analyzed (Participants) | 15 | 15 | 11 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.47 (6.13) | 66.53 (6.74) | 71.73 (5.68) | 67.24 (5.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 6 | 27
  Male | 4 | 5 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 13 | 15 | 10 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 12 | 15 | 8 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 11 | 41
Education [Mean (Standard Deviation); unit: years] | 17.83 (2.91) | 17.33 (3.21) | 16.82 (3.68) | 17.46 (6.41)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline: Memory Cognitive Domain Assessed by Montreal Cognitive Test (MoCA)
Description: To investigate the short-term effects of dental intervention on cognition, especially the memory domain of Montreal Cognitive assessment. The score ranges between 0 and 30. A score between 26 to 30 is considered to be normal. A score between 20 and 25 is for mild cognitive impairment. A score less than 20 is for Alzheimer's disease.
Time Frame: Pre and within 2 weeks post myTAP Mouth Shield intervention
Population: 41 participants consented of which 18 participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cognitively Normal Adults Group; Mild Cognitive Impairment Group; Alzheimer's Disease Group: A sample of the group will be included to investigate whether MyTAP oral airway management with a mouth shield improves sleep and cognition.
Arm/Group | Cognitively Normal Adults Group | Mild Cognitive Impairment Group | Alzheimer's Disease Group
Number analyzed (Participants) | 7 | 7 | 6
score on a scale | 28.60 (1.52) | 26.4 (1.52) | 20.6 (1.95)
Statistical Analysis 1: Comparison: Cognitively Normal Adults Group; Test type: Superiority; p = 0.05, Regression, Linear; Mean Difference (Final Values) = 2.2
Statistical Analysis 2: Comparison: Mild Cognitive Impairment Group; Test type: Superiority; p = 0.20, Regression, Linear; Mean Difference (Final Values) = 1.57
Statistical Analysis 3: Comparison: Alzheimer's Disease Group; Test type: Superiority; p = 0.642, Regression, Linear; Mean Difference (Final Values) = 0.2

ADVERSE EVENTS:
Time Frame: In period 1, the procedures administered carried minimal risk, henceforth no adverse events were noted. The subjects were followed for a period of 1 month during the assessments. In period 2, subjects were only followed during the period of interventions i.e., 6 weeks but not later than the time provided.
Description: It does not deviate from the definition mentioned in the clinical trials.gov
Groups:
- Brain Energy Metabolism and Sleep on Cognition: In the period -1 of the study, the investigator will be investigating the basic science of the relationship of sleep abnormalities, genes, brain energy metabolites variables with cognitive performance in three cohorts: cognitively normal adults, mild cognitive impairment, and Alzheimer's disease between the age of 55-85 years.
- myTAP Mouth Shield - Intervention to Improve Sleep and Cognition: To investigate if MyTAP oral airway management with mouth shield will improve sleep and cognition in three cohorts: cognitively healthy adults, mild cognitive impairment, and Alzheimer's disease between the age of 55-85 years.
  MyTAP oral appliance plus mouth shield: The midline traction oral appliance (MyTAP, AMI Inc., Dallas, Texas) is currently marketed as a medical device to treat snoring and obstructive sleep apnea and is FDA cleared will be used only in period -2 of the study. period -1 doesn't include any intervention.
Arm/Group | Brain Energy Metabolism and Sleep on Cognition | myTAP Mouth Shield - Intervention to Improve Sleep and Cognition
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/18
Other Adverse Events (participants affected / at risk) | 0/41 | 0/18

LIMITATIONS AND CAVEATS:
As covid situation started in 2019 and into 2020, the study was terminated earlier than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03929302/Prot_SAP_001.pdf